CLINICAL TRIAL: NCT05859321
Title: Effects of Virtual Reality on Pain, Functional Disability and Fear Avoidance Belief in Patients With Chronic Low Back Pain
Brief Title: Virtual Reality Based Physical Therapy for Patients With Lower Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Mwaqarafzal, Assistant Professor, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-UOL-FAHS/696-IV/2020
Record Dates: First submitted 2023-04-18; First posted 2023-05-15 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Chronic Low-back Pain
Keywords: low back pain; chronic low back pain; virtual reality
MeSH Terms: conditions — Low Back Pain | interventions — Exergaming; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality (Experimental): virtual reality exercises will be administered along with routine physiotherapy
  Interventions: Other: Virtual reality Exercises
- Routine Physiotherapy (treatment as usual) (Active Comparator): transcutaneous electrical nerve stimulation,Heat Therapy, Stretching and strengthening exercises with Cycling will be administered
  Interventions: Other: Routine Physiotherapy

INTERVENTIONS:
Other: Virtual reality Exercises — Virtual reality exercises along with transcutaneous electrical nerve stimulation, Heat Therapy and Stretching and strengthening exercises
  Arms: virtual reality
Other: Routine Physiotherapy — transcutaneous electrical nerve stimulation, Heat Therapy and Stretching and strengthening exercises
  Other Names: treatment as usual
  Arms: Routine Physiotherapy (treatment as usual)

SUMMARY:
The goal of this clinical trial is to compare chronic low back patients. The main question[s] it aims to answer are:

* pain and disability
* fear avoidance belief Participants will perform virtual reality exercises
* virtual reality based exercises
* Routine Physical Therapy To Compare routine physical therapy treatment in addition to virtual reality to see effects on pain, functional disability and fear avoidance belief

ELIGIBILITY:
Inclusion Criteria:

* Low back pain that persists for more than 12 weeks
* Non-radiating low back pain
* Mechanical low back pain
* Both Gender

Exclusion Criteria:

* trauma or fracture of the spine
* any cardiac disease
* any systematic disease
* history of any neurological diseases such as Parkinson's disease, stroke and epilepsy
* patient on corticosteroid or anticoagulants
* history of any Drug abuse
* any Congenital deformity
* Virtual reality games phobia
* Pregnant female

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-05 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | at baseline
  The Numeric Pain Rating Scale (NPRS) is a unidimensional measure of pain intensity in individuals,including those with chronic pain. Minimum socre is 0 out of 10 and Maximum 10, out of 10. Zero Indicates no pain and 10 indicates severe maximum pain.
Functional disability | at baseline
  Back pain functional scale (BPFS) is a standardized subjective assessment questionnaire that is used as Outcome tool to assess functional disability in acute and sub-acute low back pain.Minimum score is 0 out of 60 and 60 is maximum score. Zero score indicates unable to perform any functional activities and 60 indicates able to perfrom all functional activities.
Pain Intensity | at 4th week
  The Numeric Pain Rating Scale (NPRS) is a unidimensional measure of pain intensity in individuals,including those with chronic pain. Minimum socre is 0 out of 10 and Maximum 10, out of 10. Zero Indicates no pain and 10 indicates severe maximum pain.
Pain intensity | at 8th week
  The Numeric Pain Rating Scale (NPRS) is a unidimensional measure of pain intensity in individuals,including those with chronic pain. Minimum socre is 0 out of 10 and Maximum 10, out of 10. Zero Indicates no pain and 10 indicates severe maximum pain.
Functional Disability | 4th week
  Back pain functional scale (BPFS) is a standardized subjective assessment questionnaire that is used as Outcome tool to assess functional disability in acute and sub-acute low back pain.Minimum score is 0 out of 60 and 60 is maximum score. Zero score indicates unable to perform any functional activities and 60 indicates able to perfrom all functional activities.
Functional Disability | 8th week
  Back pain functional scale (BPFS) is a standardized subjective assessment questionnaire that is used as Outcome tool to assess functional disability in acute and sub-acute low back pain.Minimum score is 0 out of 60 and 60 is maximum score. Zero score indicates unable to perform any functional activities and 60 indicates able to perfrom all functional activities.

SECONDARY OUTCOMES:
Fear avoidance belief | at baseline
  Fear avoidance belief questionnaire FABQ) is a questionnaire based on the fear-avoidance model of exaggerated pain perception. The FABQ measures patient's fear of pain and consequent avoidance of physical activity (PA) because of their fear.There is a maximum score of 96. A higher score indicates more strongly held fear avoidance beliefs. There are two subscales within the FABQ; the work subscale (FABQw) with 7 questions (maximum score of 42) and the physical activity subscale (FABQpa) with 4 questions (maximum score of 24)
Range of motion | Change in range of motion score will be measured at baseline, at 8th week
  Inclinometer (minimum range of motion zero and maximum 50).
Fear avoidance belief | 4th week
  Fear avoidance belief questionnaire FABQ) is a questionnaire based on the fear-avoidance model of exaggerated pain perception. The FABQ measures patient's fear of pain and consequent avoidance of physical activity (PA) because of their fear.There is a maximum score of 96. A higher score indicates more strongly held fear avoidance beliefs. There are two subscales within the FABQ; the work subscale (FABQw) with 7 questions (maximum score of 42) and the physical activity subscale (FABQpa) with 4 questions (maximum score of 24)
Fear avoidance belief | 8th week
  Fear avoidance belief questionnaire FABQ) is a questionnaire based on the fear-avoidance model of exaggerated pain perception. The FABQ measures patient's fear of pain and consequent avoidance of physical activity (PA) because of their fear.There is a maximum score of 96. A higher score indicates more strongly held fear avoidance beliefs. There are two subscales within the FABQ; the work subscale (FABQw) with 7 questions (maximum score of 42) and the physical activity subscale (FABQpa) with 4 questions (maximum score of 24)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP, ICF